CLINICAL TRIAL: NCT00355979
Title: Randomized Trial of Intragastric Balloon and Pharmacotherapy for Non-Morbid Obesity
Brief Title: Comparative Study of Intragastric Balloon and Pharmacotherapy for Non-Morbid Obesity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2006.084
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-07

CONDITIONS: Obesity
Keywords: Obesity, intragastric balloon, Pharmacotherapy
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Device: intragastric balloon

SUMMARY:
To evaluate and compare the effectiveness of intragastric balloon and Sibutramine (Reductil®) in the treating of non-morbid obese in a randomized controlled manner

DETAILED DESCRIPTION:
Obesity is a chronic devastating disease and is becoming a major health and socioeconomic issue worldwide. Obesity significantly exacerbates many other chronic illnesses and increases mortality and morbidities of patients.1-2 Although the situation in Asians is less apparent and critical than in Caucasians, the problem is emerging rapidly. In Hong Kong, there are approximately 29% of adults classified as obese according WHO Asian criteria 3 and there is an increasing demand for obesity treatment in Asia-Pacific region.4 The first practical aim of treating obesity nowadays should focus on a sustained body weight loss of 10-15% to alleviate obesity-related illnesses such as hypertension, diabetes and obstructive sleep apnoea.

Intragastric balloon (IGB) was initially developed from observing the effects naturally caused by bezoars and the first documentation in human use was reported in 1982.5 However, earlier balloon designs were plagued by high balloon failure rates and serious complications.6-8 Since then, balloon design has undergone several major modifications in terms of material, shape and filling substances. The newer design of balloon (Bioenterics® Intragastric Balloon (BIB®) system) was introduced in 1999 9 and has undergone extensive evaluation recently in Europe with promising results.10-11 It is placed inside the stomach endoscopically for a maximum of 180 days to decrease stomach capacity and gastric emptying. It facilitates patient's compliance to the restricted diet prescribed and together with increasing level of physical activities, most reports have shown moderate body weight loss of 15 % or more.10--12 More importantly, the newer design balloon (BIB) is more reliable and predictable. The reported premature balloon rupture and serious complication is rare if it is removed within the recommended period and followed up carefully by a dedicated obesity team in a multidisciplinary approach.10-12 Sibutramine (Reductil®) is a serotonin and noradrenaline reuptake inhibitor and is one of the FDA approved weight reduction pharmacotherapy. Its central action on neurotransmitters causes an enhancement of satiety (fullness) after eating. In addition, it causes sympathetically mediated thermogenesis, which prevent the reduction in basal metabolic rate (BMR) normally seen in individual on restricted diet and thereby effectively increases resting energy consumption and promotes weight loss. A combination of sibutramine and lifestyle modification program has been shown up to 10 % of body weight loss while intragastric balloon and sibutramine are the two most commonly used non-surgical method for weight reduction. There is lack of randomized controlled trial in comparing these two methods in the treatment of obesity. Since these two types of therapy are most efficient in non-morbid obese patients, we are designing a trial to compare the effect of the two different weight reduction therapies in this group of patients in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60
2. BMI 27-35
3. Agree to undergo invasive weight reduction therapy and intensive follow-up
4. No history of weight reduction for >5% of BW for the past 6 months

Exclusion Criteria:

1. Coronary heart disease
2. Un-controlled hypertension (160/90 mmHg)
3. unstable cardiovascular disease
4. unstable cerebrovascular disease
5. Renal disease
6. Liver disease

9) Diabetes Mellitus 10) Eating disorder 11) Psychiatric illness 12) Pregnant or breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2006-03; Study Completion 2008-03

PRIMARY OUTCOMES:
Body weight loss in terms of % of body weight and BMI loss at 6-month and 1 year.

SECONDARY OUTCOMES:
Regain of weight after treatment, complications and compliance of treatment, change of satiety level and calorie intake during and after treatment, quality of life, change in hormonal profile and patient's satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred LM Mui, FRCS, Principal Investigator — The Chinese University of Hong Kong, Hong Kong ,China
Locations (1):
- The Chinese University of Hong Kong, Department of Surgery, Hong Kong, Hong Kong, China